CLINICAL TRIAL: NCT04363671
Title: Qualitative Study of the Experience of Adolescents and Health Professionals Faced With the Necessity for Changing to Remote Care During the COVID-19 Outbreak Quarantine
Brief Title: Adolescents and Health Professionals Faced With the Necessity for Changing to Remote Care During the COVID-19 Outbreak Quarantine (AdoPro-Cov19)
Acronym: AdoPro-Cov19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hôpital Cochin (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Carretier Emilie, MD Psychiatrist, Hôpital Cochin
Other Study IDs: P20-670
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Remote Consultation; Covid-19
Keywords: Qualitative research; Adolescent; Health personnel attitude; Coronavirus; Quanrantine
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Maison des Adolescents (MDA) at Cochin Hospital (Paris) is a multidisciplinary service which welcomes adolescents in three different units: consultation, day care and hospitalization. However, the epidemic of coronavirus (COVID-19) in March 2020 which imposed the extreme limitation of contacts and then the confinement of the entire population, required urgent adaptation of care practices. Teleconsultation quickly became essential for most consultations (psychiatrists, psychologists, nurses, but also pediatricians and somatic physicians). In day hospital, daily reception could not be carried out, therapeutic workshops, family interviews, or speaking groups were organized remotely. In hospital unit, the interruption of visits required the organization of remote interviews with families. Far from the comfort of an organized and structured telepsychiatry, the use of videoconferencing was done in an emergency and without preparation. The objective is to explore the experience of adolescents, doctors and psychologists regarding emergency changes in the methods of their follow-up by setting up teleconsultation in the context of the COVID-19 epidemic.

DETAILED DESCRIPTION:
The study will be monocentric, exploratory, and qualitative based on the Interpretative Phenomenological Analysis. 15 adolescents followed in consultation, day hospital or full hospitalization and 15 health professionals working at the Maison des Adolescents will be included. Semi-structured interviews will be carried out by a psychiatrist, based on flexible and evolving interview guides. Qualitative analysis of adolescents and therapists' interviews will allow to explore the experience of teleconsultation by each group of participants and to inform about the advantages and limits of a teleconsultation device in adolescent care.

ELIGIBILITY:
Inclusion Criteria:

* adolescents aged between 11 and 20 years who benefit from follow-up in the structure (at least two face-to-face consultations before setting up teleconsultations) and for whom their follow-up had to be changed urgently in the form of teleconsultation from March 2020 as part of the COVID-19 epidemic. Adolescents will be included in the various consultation, day hospitalization and full hospitalization units. The pathologies will be varied so as to cover different situations and experiences: eating disorders, mood disorders, personality disorders, anxiety disorders, or even chronic somatic illness.
* health professionals working at the Maison des Adolescents at the time of the epidemic, from different specialties (psychiatrists, pediatricians, psychologists, nurses, etc.) and units (consultations, day hospitalization, full hospitalization).

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 15 adolescents followed in consultation, day hospital or full hospitalization and 15 health professionals working at the MDA during the COVID-19 epidemic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Exploration of themes emerging from analysis of the content of the interview with the adolescents and therapists | six months
  To describe the experience of reorganization of care during the COVID-19 epidemic and acceptability of teleconsultation for the adolescents and the therapists.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Carretier, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Maison de Solenn, Cochin Hospital, Paris, France